CLINICAL TRIAL: NCT00478894
Title: Multicenter Orthopaedic Outcomes Network (MOON) Anterior Cruciate Ligament (ACL) Reconstruction (ACLR): Onsite Follow-up
Brief Title: Multicenter Orthopaedic Outcomes Network (MOON) ACL Reconstruction (ACLR): Onsite Follow-up
Acronym: MOON-Onsite
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Kurt P. Spindler, Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 070264; 5R01AR053684 (NIH)
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Rupture of Anterior Cruciate Ligament; Osteoarthritis
Keywords: Anterior cruciate ligament / injuries; Anterior cruciate ligament / surgery; knee injuries / surgery; outcomes research; prospective studies; osteoarthritis
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis; Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this study we will examine patients who have undergone unilateral ACL reconstruction surgery to determine which structural and functional characteristics of the knee two and ten years post reconstruction surgery, aspects of the original injury and repair, and patient characteristics are risk factors for osteoarthritis after ACL reconstruction surgery.

DETAILED DESCRIPTION:
The purpose of this study is identify risk factors for signs and symptoms of osteoarthritis two and ten year post ACL reconstruction from information available at the time of surgery; including patient characteristics (age, gender, body mass index (BMI), activity level, clinical knee alignment), their injuries ("pop" heard at the time of injury, concurrent meniscus, articular cartilage, and collateral ligament injuries), and treatment decisions made during the initial surgery (e.g. meniscus and articular cartilage treatments.)

Primary outcome measures will be the Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain and stiffness subscales and joint space width measured on weight-bearing radiographs.

Secondary outcome measures will include the knee related quality of life subscale of the Knee Injury and Osteoarthritis Score (KOOS) and Kellgren-Lawrence grading from weight-bearing radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Had primary unilateral ACL reconstruction performed by Dr. Kurt Spindler (Vanderbilt University), Dr. Christopher Kaeding (The Ohio State University), Dr. Rick Parker (Cleveland Clinic), Dr. Jack Andrish (Cleveland Clinic), Dr. Rick Wright (Washington University in St. Louis), or Dr. Matthew Matava (Washington University in St. Louis)
* 14-55 years of age at the time of follow-up

Exclusion Criteria:

* less than 14 years or greater than 55 years
* non-active or unable to participate for health reasons

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants enrolled in the Multicenter Orthopaedic Outcomes Network cohort by one of three surgeons and meeting eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2007-08; Primary Completion 2025-12 (Actual); Study Completion 2025-12 (Actual)

PRIMARY OUTCOMES:
Side to side knee joint space difference as seen on x-ray | 2-20 years post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kurt P Spindler, M.D., Principal Investigator — Cleveland Clinic / Vanderbilt University
Locations (4):
- United States (4):
  - Washington University in St. Louis, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Result] Reinke EK, Spindler KP, Lorring D, Jones MH, Schmitz L, Flanigan DC, An AQ, Quiram AR, Preston E, Martin M, Schroeder B, Parker RD, Kaeding CC, Borzi L, Pedroza A, Huston LJ, Harrell FE Jr, Dunn WR. Hop tests correlate with IKDC and KOOS at minimum of 2 years after primary ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2011 Nov;19(11):1806-16. doi: 10.1007/s00167-011-1473-5. Epub 2011 Mar 29. PMID 21445595
- [Derived] Ramkumar PN, Tariq MB; MOON Knee Group; Amendola A, Andrish JT, Brophy RH, Dunn WR, Flanigan DC, Huston LJ, Jones MH, Kaeding CC, Kattan MW, Marx RG, Matava MJ, McCarty EC, Parker RD, Vidal AF, Wolcott ML, Wolf BR, Wright RW, Spindler KP. Risk Factors for Loss to Follow-up in 3202 Patients at 2 Years After Anterior Cruciate Ligament Reconstruction: Implications for Identifying Health Disparities in the MOON Prospective Cohort Study. Am J Sports Med. 2019 Nov;47(13):3173-3180. doi: 10.1177/0363546519876925. Epub 2019 Oct 7. PMID 31589465
- [Derived] Jacobs CA, Peabody MR, Lattermann C, Vega JF, Huston LJ, Spindler KP; MOON Knee Group; Amendola A, Andrish JT, Brophy RH, Dunn WR, Flanigan DC, Jones MH, Kaeding CC, Marx RG, Matava MJ, McCarty EC, Parker RD, Reinke EK, Wolcott ML, Wolf BR, Wright RW, Vidal AF. Development of the KOOSglobal Platform to Measure Patient-Reported Outcomes After Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2018 Oct;46(12):2915-2921. doi: 10.1177/0363546518789619. Epub 2018 Aug 3. PMID 30074823